CLINICAL TRIAL: NCT03599336
Title: Reverse Total Shoulder Arthroplasty Versus Nonoperative Treatment of 3 & 4-Part Proximal Humerus Fractures
Brief Title: RSA vs. Nonop for 3 & 4-Part Proximal Humerus Fractures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slower than expected enrollment.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jonathan D. Barlow, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-002097
Record Dates: First submitted 2018-06-30; First posted 2018-07-26 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Humerus Fracture; Humerus; Shoulder Fractures; Shoulder Arthropathy Associated With Other Conditions; Arthropathy Shoulder; Shoulder Injury; Arthropathy
MeSH Terms: conditions — Humeral Fractures; Shoulder Fractures; Shoulder Injuries; Joint Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nonoperative Treatment (Other): Subjects will have nonoperative treatment to treat proximal humerus fracture that is broken into 3 or 4 parts.
  Interventions: Other: Nonoperative Treatment
- Operative Course for rTSA (Other): Subjects will have shoulder replacement surgery to treat proximal humerus fracture that is broken into 3 or 4 parts.
  Interventions: Procedure: Reverse Total Shoulder Arthroplasty (rTSA)

INTERVENTIONS:
Procedure: Reverse Total Shoulder Arthroplasty (rTSA) — Surgical management will include placement of fracture specific, cemented reverse total shoulder arthroplasty components as per standard surgical care and routine postoperative rehabilitation.
  Arms: Operative Course for rTSA
Other: Nonoperative Treatment — Subjects allocated to the nonoperative treatment arm will maintain sling immobilization for 3 weeks. The sling will be removed for elbow, wrist and hand range of motion (ROM), hygiene, and dressing only. At 3 weeks passive ROM in external rotation (ER) and forward elevation (FE) will be added. At 6 weeks from injury, the sling will be removed and stretching in all planes will be allowed. Use of the arm will be up to a fork/knife/toothbrush only. At 3 months from injury, strengthening will be added. Supervised physical therapy will be offered to patients for use at their discretion, as is current practice.
  Arms: Nonoperative Treatment

SUMMARY:
There is currently no consensus amongst orthopedic specialists on the best way to treat 3- and 4-part proximal humerus fractures. No surgery and surgery with a type of shoulder replacement called a reverse total shoulder arthroplasty are two options that many orthopedists use. This study is being performed to evaluate the differences in short- and long-term pain and functional outcomes between patients who are treated with these two different options.

ELIGIBILITY:
Inclusion criteria

* Displaced 3- and 4-part proximal humerus fractures.
* Age greater than or equal to 65 years old.

Exclusion Criteria

* Less than 65 years old.
* Medical comorbidities precluding surgical treatment or anesthesia
* Dementia or inability to provide adequate follow up.
* Pathologic fractures
* Open fractures
* Associated injuries: fracture dislocations, multiple or complex injuries of the ipsilateral limb, complete brachial plexopathy, vascular injury and polytrauma.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2020-10-29 (Actual)

PRIMARY OUTCOMES:
Function as described by ASES score at 1 year follow-up. | 2 year follow-up
  The American Shoulder and Elbow Surgeons (ASES) score is a well-validated, patient-reported outcome measure used by shoulder and elbow surgeons. The score ranges from 0-100 with 100 signifying the best outcome. Half of the score correlates to pain and half to function, both on a 0-50 scale where higher is again considered a better outcome. The pain portion is tabulated by taking the patient's response on a visual analogue scale (0 to 10 scale where 0 represent no pain and 10 represents worst pain imaginable), subtracting it from 10, and then multiplying by 5. The function score is tabulated by taking the patient's response on 10 questions rated on an ordinal scale from 0-3 and then multiplying the cumulative score by 5/3.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D Barlow, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials